CLINICAL TRIAL: NCT01658098
Title: Prevalence of Postpartum Depression in the Jose E. Gonzalez Hospital, Using the Edinburgh Postpartum Depression Scale
Brief Title: Prevalence of Postpartum Depression in Hospital Jose E. Gonzalez
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hospital Universitario Dr. Jose E. Gonzalez (Other)
Responsible Party: Principal Investigator, Dr Edgar Alejandro Tamez Cristerna, principal investigator, Hospital Universitario Dr. Jose E. Gonzalez
Other Study IDs: etamez
Record Dates: First submitted 2012-07-30; First posted 2012-08-06 (Estimated); Last update posted 2012-08-06 (Estimated); Status verified 2012-07

CONDITIONS: Postpartum Depression
Keywords: postpartum; depression; edinburgh postpartum depression scale; mexican population
MeSH Terms: conditions — Depression, Postpartum; Depression

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- 4-6 weeks after delivery: all patients on their 4th-6th weeks after delivery
  Interventions: Behavioral: edinburgh postpartum depression scale questionary

INTERVENTIONS:
Behavioral: edinburgh postpartum depression scale questionary — the investigators will apply the qusetionary one time only in the period of time described previously

SUMMARY:
This research will use the Edinburgh Scale Of Post partum depression to evaluate patients during their 4th to 6th after delivery, and the investigators will compare the results with those found in other countries with population with similar characteristics as ours

ELIGIBILITY:
Inclusion Criteria:

* patients on their 4th -6th week after delivery, who gave birth in our institution

Exclusion Criteria:

* patients with previous diagnosis of psychiatric pathology

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 348 patients on their 4th-6th week after delivery
Sampling Method: Probability Sample
Enrollment: 348 (Estimated)
Dates: Start 2012-09; Primary Completion 2012-11 (Estimated); Study Completion 2013-02 (Estimated)

PRIMARY OUTCOMES:
presence of postpartum depression | 2 months

SECONDARY OUTCOMES:
sociodemographic characteristics | 2 months
  age
sociodemographic characteristics | 2 month
  level of education
obstetrical background | 2 month
  number of pregnancies
medical background | 2 month
  comorbid ities

CONTACTS AND LOCATIONS:
Overall Officials: Emilio Treviño, specialist, Study Director — Consejo mexicano de ginecologia y obstetricia
Locations (1):
- Hospital Universitario Dr Jose E. Gonzalez, Monterrey, Nuevo León, Mexico

REFERENCES:
- [Background] Dennis CL. Can we identify mothers at risk for postpartum depression in the immediate postpartum period using the Edinburgh Postnatal Depression Scale? J Affect Disord. 2004 Feb;78(2):163-9. doi: 10.1016/s0165-0327(02)00299-9. PMID 14706728
- [Background] Yang SN, Shen LJ, Ping T, Wang YC, Chien CW. The delivery mode and seasonal variation are associated with the development of postpartum depression. J Affect Disord. 2011 Jul;132(1-2):158-64. doi: 10.1016/j.jad.2011.02.009. Epub 2011 Mar 4. PMID 21377210
- [Background] Petrosyan D, Armenian HK, Arzoumanian K. Interaction of maternal age and mode of delivery in the development of postpartum depression in Yerevan, Armenia. J Affect Disord. 2011 Dec;135(1-3):77-81. doi: 10.1016/j.jad.2011.06.061. Epub 2011 Aug 10. PMID 21835474
- [Background] Xie RH, He G, Liu A, Bradwejn J, Walker M, Wen SW. Fetal gender and postpartum depression in a cohort of Chinese women. Soc Sci Med. 2007 Aug;65(4):680-4. doi: 10.1016/j.socscimed.2007.04.003. Epub 2007 May 15. PMID 17507127
- [Background] Pearlstein T, Howard M, Salisbury A, Zlotnick C. Postpartum depression. Am J Obstet Gynecol. 2009 Apr;200(4):357-64. doi: 10.1016/j.ajog.2008.11.033. PMID 19318144
- [Background] Jadresic E, Nguyen DN, Halbreich U. What does Chilean research tell us about postpartum depression (PPD)? J Affect Disord. 2007 Sep;102(1-3):237-43. doi: 10.1016/j.jad.2006.09.032. Epub 2006 Nov 27. PMID 17125843
- [Background] Affonso DD, De AK, Horowitz JA, Mayberry LJ. An international study exploring levels of postpartum depressive symptomatology. J Psychosom Res. 2000 Sep;49(3):207-16. doi: 10.1016/s0022-3999(00)00176-8. PMID 11110992
- [Background] Sylven SM, Papadopoulos FC, Olovsson M, Ekselius L, Poromaa IS, Skalkidou A. Seasonality patterns in postpartum depression. Am J Obstet Gynecol. 2011 May;204(5):413.e1-6. doi: 10.1016/j.ajog.2011.01.022. Epub 2011 Mar 24. PMID 21439544
- [Background] Halbreich U, Karkun S. Cross-cultural and social diversity of prevalence of postpartum depression and depressive symptoms. J Affect Disord. 2006 Apr;91(2-3):97-111. doi: 10.1016/j.jad.2005.12.051. Epub 2006 Feb 7. PMID 16466664
- [Background] Miyake Y, Tanaka K, Sasaki S, Hirota Y. Employment, income, and education and risk of postpartum depression: the Osaka Maternal and Child Health Study. J Affect Disord. 2011 Apr;130(1-2):133-7. doi: 10.1016/j.jad.2010.10.024. Epub 2010 Nov 4. PMID 21055825
- [Background] Latorre-Latorre JF, Contreras-Pezzotti LM, Herran-Falla OF. [Postnatal depression in a Colombian city. Risk factors]. Aten Primaria. 2006 Apr 15;37(6):332-8. doi: 10.1157/13086714. Spanish. PMID 16733006
- [Background] Delatte R, Cao H, Meltzer-Brody S, Menard MK. Universal screening for postpartum depression: an inquiry into provider attitudes and practice. Am J Obstet Gynecol. 2009 May;200(5):e63-4. doi: 10.1016/j.ajog.2008.12.022. Epub 2009 Mar 14. PMID 19285644
- [Background] Hewitt C, Gilbody S, Brealey S, Paulden M, Palmer S, Mann R, Green J, Morrell J, Barkham M, Light K, Richards D. Methods to identify postnatal depression in primary care: an integrated evidence synthesis and value of information analysis. Health Technol Assess. 2009 Jul;13(36):1-145, 147-230. doi: 10.3310/hta13360. PMID 19624978
- [Background] Jadresic E, Araya R, Jara C. Validation of the Edinburgh Postnatal Depression Scale (EPDS) in Chilean postpartum women. J Psychosom Obstet Gynaecol. 1995 Dec;16(4):187-91. doi: 10.3109/01674829509024468. PMID 8748993
- [Background] Castanon S C, Pinto L J. [Use of the Edinburgh Postnatal Depression Scale to detect postpartum depression]. Rev Med Chil. 2008 Jul;136(7):851-8. Epub 2008 Sep 4. Spanish. PMID 18949160
- [Background] Gibson J, McKenzie-McHarg K, Shakespeare J, Price J, Gray R. A systematic review of studies validating the Edinburgh Postnatal Depression Scale in antepartum and postpartum women. Acta Psychiatr Scand. 2009 May;119(5):350-64. doi: 10.1111/j.1600-0447.2009.01363.x. Epub 2009 Mar 2. PMID 19298573